CLINICAL TRIAL: NCT00004173
Title: A Phase I Study of Oxaliplatin in Combination With Paclitaxel
Brief Title: Oxaliplatin and Paclitaxel in Treating Patients With Metastatic or Unresectable Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: OSU-99H0284; CDR0000067419 (Registry Identifier: PDQ (Physician Data Query)); NCI-T99-0017
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2003-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Oxaliplatin; Paclitaxel

INTERVENTIONS:
Drug: oxaliplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of oxaliplatin and paclitaxel in treating patients who have metastatic or unresectable cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of oxaliplatin and paclitaxel in patients with metastatic or unresectable cancer.
* Determine the qualitative and quantitative toxicities of this regimen in these patients.
* Determine the therapeutic response to this regimen in these patients.
* Determine the relationship between the pharmacokinetics of this regimen and toxicity and response in these patients.
* Determine the effects of oxaliplatin on peripheral blood cells and correlate this to pharmacokinetics, toxicity, and response in these patients.

OUTLINE: This is a dose escalation study.

Patients receive oxaliplatin IV over 2 hours followed by paclitaxel IV over 1 hour weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin and paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic or unresectable malignancy for which standard curative or palliative measures do not exist or are no longer effective
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2
* Karnofsky 50-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3000/mm^3
* Absolute neutrophil count at least 1500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* SGOT/SGPT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No neuropathy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No allergy to platinum compounds or antiemetics
* No uncontrolled concurrent illness
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 2 prior chemotherapy regimens
* No prior oxaliplatin or paclitaxel
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow

Surgery:

* Not specified

Other:

* No other concurrent investigational agents
* No concurrent antiretroviral therapy for HIV (HAART)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Eric H. Kraut, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio, United States